CLINICAL TRIAL: NCT00699660
Title: Enhancing Equitable and Effective PTSD Disability Assessment
Brief Title: Enhancing Equitable and Effective (E-3) Post Traumatic Stress Disorder (PTSD) Disability Assessment
Acronym: E-3PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SDR 06-331
Record Dates: First submitted 2008-06-12; First posted 2008-06-18 (Estimated); Results first posted 2014-10-16 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-07

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Disability Examination; Clinician Administered PTSD Scale; Quality of Care
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CAPS/WHODAS (Experimental): PTSD assessed using Clinical Assessment of PTSD Symptoms (CAPS) and WHODAS functional impairment structured evidence-based interview
  Interventions: Behavioral: CAPS/WHODAS
- Nonstructured Interview (Active Comparator): Usual clinical interview to assess PTSD, without CAPS or WHODAS
  Interventions: Behavioral: Nonstructured Interview

INTERVENTIONS:
Behavioral: CAPS/WHODAS — CAPS/WHODAS structured clinical PTSD interview
  Arms: CAPS/WHODAS
Behavioral: Nonstructured Interview — Usual PTSD clinical PTSD interview, not CAPS or SCID
  Other Names: Usual Clinical Interview
  Arms: Nonstructured Interview

SUMMARY:
This project evaluated the impact of semi-structured, standardized interviews on the initial PTSD C&P on the examination.

DETAILED DESCRIPTION:
Our objective is to compare the process and outcomes of C&P exams for PTSD conducted with CAPS and WHODAS-II interviews versus the PTSD exams conducted without the CAPS and WHODAS-II interviews. This project will conduct a randomized controlled trial on 688 veterans to evaluate the effects of the CAPS/WHODAS instruments on the initial PTSD C&P examination process. Study outcomes include variation in assessing the DSM-IV components of PTSD, diagnostic accuracy, veteran perception of the exam process, VBA rater utility and resource utilization. This project will 1) demonstrate the feasibility of conducting program evaluation and intervention studies on the PTSD C&P examination process, 2) develop research tools, instruments and methods for C&P evaluation, 3) provide data on the value-added contribution of CAPS and WHODAS-II to the PTSD assessment process and examination report, and 4) inform the business case of utilizing the CAPS and WHODAS-II in the PTSD C&P process. The ultimate aim is to improve the reproducibility, consistency and validity of the PTSD examination process while maintaining a level of efficiency and cost restraint that provides veterans with an exam process that is fair, accurate and equitable across VHA.

ELIGIBILITY:
Inclusion Criteria:

1. Veterans referred to VHA for an Initial PTSD Compensation and Pension Examination
2. Informed consent

Exclusion Criteria:

1. Mentally impaired, not able to give informed consent
2. English speaking

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2009-05; Primary Completion 2010-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Speroff, PhD, Principal Investigator — Tennessee Valley Healthcare System Nashville Campus, Nashville, TN
Locations (11):
- United States (11):
  - Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR, North Little Rock, Arkansas
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - Southeast Louisiana Veterans Health Care System, New Orleans, LA, New Orleans, Louisiana
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - John D. Dingell VA Medical Center, Detroit, MI, Detroit, Michigan
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - New Mexico VA Health Care System, Albuquerque, NM, Albuquerque, New Mexico
  - Memphis VA Medical Center, Memphis, TN, Memphis, Tennessee
  - Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee
  - Clement J. Zablocki VA Medical Center, Milwaukee, WI, Milwaukee, Wisconsin

REFERENCES:
- [Result] Rosen MI, Afshartous D, Marx BP. Did microinsults and microaggressions play a role?: in reply. Psychiatr Serv. 2013 Jul 1;64(7):713. doi: 10.1176/appi.ps.640703. No abstract available. PMID 23821175
- [Result] Rosen MI, Afshartous DR, Nwosu S, Scott MC, Jackson JC, Marx BP, Murdoch M, Sinnott PL, Speroff T. Racial differences in veterans' satisfaction with examination of disability from posttraumatic stress disorder. Psychiatr Serv. 2013 Apr 1;64(4):354-9. doi: 10.1176/appi.ps.201100526. PMID 23318842
- [Result] Speroff T, Sinnott PL, Marx B, Owen RR, Jackson JC, Greevy R, Sayer N, Murdoch M, Shane AC, Smith J, Alvarez J, Nwosu SK, Keane T, Weathers F, Schnurr PP, Friedman MJ. Impact of evidence-based standardized assessment on the disability clinical interview for diagnosis of service-connected PTSD: a cluster-randomized trial. J Trauma Stress. 2012 Dec;25(6):607-15. doi: 10.1002/jts.21759. PMID 23225029
- [Result] Marx BP, Jackson JC, Schnuff PP, Murdoch M, Sayer NA, Keane TM, Friedman MJ, Greevy RA, Owen RR, Sinnott PL, Speroff T. The reality of malingered PTSD among Veterans: Reply to McNally and Frueh. Journal of traumatic stress. 2012 Aug 1; 25(4):457-60.
- [Result] Jackson JC, Sinnott PL, Marx BP, Murdoch M, Sayer NA, Alvarez JM, Greevy RA, Schnurr PP, Friedman MJ, Shane AC, Owen RR, Keane TM, Speroff T. Variation in practices and attitudes of clinicians assessing PTSD-related disability among veterans. J Trauma Stress. 2011 Oct;24(5):609-13. doi: 10.1002/jts.20688. Epub 2011 Sep 12. PMID 21913226
- [Result] Marx BP, Marshall PJ, Castro F. The moderating effects of stimulus valence and arousal on memory suppression. Emotion. 2008 Apr;8(2):199-207. doi: 10.1037/1528-3542.8.2.199. PMID 18410194
- [Result] Sloan DM, Marx BP, Epstein EM, Dobbs JL. Expressive writing buffers against maladaptive rumination. Emotion. 2008 Apr;8(2):302-6. doi: 10.1037/1528-3542.8.2.302. PMID 18410204

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: PTSD interview using CAPS and WHODAS
  Clinician Assessment of PTSD Symptoms (CAPS): CAPS/WHODAS structured clinical PTSD interview
- Arm 2: Usual PTSD interview, without CAPS or WHODAS
  Nonstructured Interview: Usual PTSD clinical PTSD interview, not CAPS or SCID
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 190 | 216
Completed | 176 | 208
Not Completed | 14 | 8
Not completed — Lost to Follow-up | 4 | 2
Not completed — missing reports and recording failures | 10 | 6

BASELINE CHARACTERISTICS:
Population: Veterans undergoing compensation and pension examination for PTSD
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 176 | 208 | 384
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [41 to 63] | 59 [41 to 62] | 59 [41 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 13 | 19
  Male | 170 | 195 | 365
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 44 | 56 | 100
  White | 103 | 124 | 227
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 29 | 28 | 57
Marital Status [Number; unit: participants]
  Married | 108 | 130 | 238
  Single | 28 | 35 | 63
  Separated | 32 | 37 | 69
  Other/Missing | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Completeness and Quality of PTSD Interview
Description: total completeness of diagnostic assessment score, range from 0 to 100% and completeness of functional assessment
Time Frame: Post-exam, same day
Measure: Mean (Standard Deviation); unit: percentage of criteria PTSD assessment
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 176 | 208
percentage of criteria PTSD assessment
  completeness of diagnostic assessment | 84.8 (17.3) | 29.8 (24.4)
  completeness of functional assessment | 76.2 (24.4) | 3.1 (7.5)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Our sample size calculation yielded 466 for a power of 0.80 to detect a 10% absolute difference in sensitivity and adjusted for intraclass correlation. The number of covariates in regression models was limited to ensure the effective sample size remained ten times greater than the degrees of freedom in the model; Test type: Superiority or Other; p < .001, Regression, Linear — Comparison of CAPS/WHODAS vs Nonstructured Interview study arms: linear and logistic mixed effects regression with clinical examiner stratified by study group as a random effect and study group as a fixed effect; Covariates included experience, use of template,tests,reviewing records,age,education, study site,reviewer, and expert reviewer by group interaction

2. Secondary Outcome: PTSD Diagnosis
Description: Number of participants who were unable to receive a conclusive clinician PTSD diagnosis for positive or negative PTSD symptoms (unable to determine clinician diagnosis).
Time Frame: Post-exam, same day
Measure: Number; unit: participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 176 | 208
participants
  Uanble to determine clinician PTSD+ diagnosis | 49 | 110
  Unable to determine PTSD- diagnosis | 14 | 73
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Superiority or Other; p < .01, Regression, Logistic

3. Secondary Outcome: Patient Satisfaction
Description: Mean score on satisfaction survey rating scale from 1 to 5 (higher)
Time Frame: post-exam, same day
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 176 | 208
units on a scale | 4.69 (.44) | 4.74 (.38)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Superiority or Other; p > .05, t-test, 2 sided — Descriptive statistics on mean and standard deviation

4. Secondary Outcome: Resource Utilization
Description: time spent administering the exam
Time Frame: same day
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 176 | 208
minutes | 216.6 (88.6) | 157.2 (63.8)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Estimates of the influence on total time and tests of statistical significance were derived from multilevel mixed-effects linear regression (xtmixed in Stata); Test type: Superiority or Other; p = .012, Regression, Linear — 0.05 level based on a two tailed test; Covariates included years of experience, use of template, use of tests, age, education, study site; Slope = 47.3, Standard Error of Mean 18.86

ADVERSE EVENTS:
Time Frame: Day of disability examination
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/176 | 0/208
Other Adverse Events (participants affected / at risk) | 0/176 | 0/208

LIMITATIONS AND CAVEATS:
Information external to interview such as psychological testing or charts were not available to the expert reviewers. Another limitation is that Veterans in our study did not undergo a concurrent, independent evaluation for assessment of PTSD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No